CLINICAL TRIAL: NCT01569776
Title: Evaluation of Hypoallergenicity of an Amino Acid-Based Infant Formula
Brief Title: Elemental Formula Hypoallergenicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09.55.PED
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Food Hypersensitivity
Keywords: Cow milk allergy; CMA
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Amino Acid formula (Experimental)
  Interventions: Other: Amino Acid formula
- Control formula (Active Comparator): Commercially available Amino Acid infant formula
  Interventions: Other: Commercially available Amino Acid Formula

INTERVENTIONS:
Other: Amino Acid formula — Amino Acid baby formula
  Arms: New Amino Acid formula
Other: Commercially available Amino Acid Formula — Hypoallergenic Baby formula
  Arms: Control formula

SUMMARY:
The primary objective of this clinical trial is to determine whether a new amino acid-based formula is hypoallergenic as defined by the American Academy of Pediatrics (2000), demonstrating that the test formula does not provoke allergenic activity in 90% of infants or children with confirmed cow's milk allergy (CMA) with 95% confidence as compared to a commercially available hypoallergenic formula.

ELIGIBILITY:
Inclusion Criteria:

* Born at term (>36 weeks gestation)
* 2 months to ≤12 years of age at enrollment
* Documented CMA within 6 months prior to enrollment
* Otherwise healthy
* Asthma, atopic dermatitis and/or rhinitis must be well-controlled, if applicable
* Expected daily intake of at least 8 oz (240ml) of the study formula during the open challenge phase
* Having obtained his/her legal representative's informed consent

Exclusion:

* Children consuming mother's milk at the time of inclusion and during the trial
* Any chromosomal or major congenital anomalies
* Any major gastrointestinal disease or abnormalities other than CMA
* Chronic medical diseases (ie seizure disorders, chronic lung disease, heart problems (heart murmurs okay)
* Immunodeficiency
* Anti-histamine use in 7 days prior to the first food challenge (eyedrops are permitted)
* Oral steroid use within 14 days prior to enrollment (intranasal and topical corticosteroid use are permitted)
* Unstable asthma
* Severe uncontrolled eczema
* Severe anaphylactic reaction to milk within the last 2 years
* Severe anaphylactic reaction to breastmilk within the last 2 years
* Subject who in the Investigator's assessment cannot be expected to adhere to the study protocol
* Currently participating in another clinical trial.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
occurrence of allergic reactions | 14 days
  occurrence of allergic reactions to double-blind placebo controlled food challenge (DBPCFC)

SECONDARY OUTCOMES:
Digestive Tolerance | one week
  gastrointestinal tolerance and formula intake recorded during the open challenge phase.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nowak-Wegrzyn, MD, Principal Investigator — Mount Sinai Department of Pediatrics
Locations (9):
- United States (9):
  - Pediatric Care Medical Group, Inc., Huntington Beach, California
  - Allergy & Asthma Medical Group and Research Center, A P.C., San Diego, California
  - Georgia Pollens Clinical Research Centers Inc., Albany, Georgia
  - Allergy & Asthma Physicians, Hinsdale, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Mount Sinai Medical Center, New York, New York
  - ENT & Allergy Associates, Newburgh, New York
  - TTS Research, Boerne, Texas
  - Clinical Research Partners, Richmond, Virginia

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765